CLINICAL TRIAL: NCT04458142
Title: Comparison of The Efficiency of Single Buccal Infiltration Versus Buccal and Intrapapillary Infiltration Using 4% Articaine During Extraction of Primary Maxillary Molar Teeth: A Randomized Controlled Trial Split Mouth Design Study
Brief Title: Efficiency of Single Buccal Infiltration Versus Buccal and Intrapapillary Infiltration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadil Ahmed Mohamed Ahmed ELSafty, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422017496954
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single buccal infiltration using 4%articaine (Experimental): Dryness the site of injection then application of topical anesthetic gel(2% benzocaine).
  Injecting by a small amount of solution in the superficial mucosa. After a few seconds, the needle was slowly advanced in the mucobuccal fold toward the apex of the molar and 1.8 ml of 4% articaine using short 30-gauge needle was slowly given.
  Subjective assessment of buccal and palatal soft tissue anesthesia will be assessed by inquiring about the area of numbness from the participant, no pain during pricking the palatal mucosa. The cases in which palatal anesthesia will not be reported by the patient will be given supplemental palatal infiltration with 0.2 to 0.3 mL articaine.
  After achieving adequate buccal and palatal tissue anesthesia, the tooth will be extracted under aspetic technique.
  Interventions: Other: Single buccal infiltration
- Buccal and intrapapillary infiltration using 4%articaine (Active Comparator): Dryness the site of injection then application of topical anesthetic gel(2% benzocaine) Injecting a small amount of solution in the superficial mucosa,then needle will slowly advanced in the mucobuccal fold toward the apex of the molar and 1.5 ml of 4% articaine was slowly given. The remaining 0.3ml solution will be given equally into the distal, mesial intrapapillary and palatal sites respectively until blanching of the palate is observed extending more than halfway along the palatal gingival margin.
  Subjective assessment of buccal and palatal soft tissue anesthesia will be assessed.
  After achieving adequate buccal and palatal tissue anesthesia, the tooth will be extracted under aspetic technique.
  Interventions: Other: Single buccal infiltration

INTERVENTIONS:
Other: Single buccal infiltration — painless technique for palatal anesthesia,single injection,single puncture given

SUMMARY:
Everyday practice in dentistry is based on giving the painless injection and achieving adequate local anesthesia. Various techniques of reducing injection pain in children can be broadly categorized as psychological and physical. The psychological approach includes behavior management techniques, physical means and other recent techniques such as computer controlled anesthesia, electronic dental anesthesia, and so forth. However, none of these techniques have been successful in eliminating pain, fear and anxiety in children.

Direct palatal injection technique is difficult to administer without significant pain or discomfort since there is little tissue space at these sites between the mucosa and the underlying periosteum. Studies conducted on indirect palatal injection technique (intrapapillary) revealed that it reduces the pain of palatal injection with the same efficacy of anesthesia during extraction.

The desirable method to evade pain during palatal injection is just not to have one.

Maxillary molars removal without palatal or multiple injections is possible due to relatively thin porous bone of posterior buccal maxilla that facilitates the diffusion of local anesthetic.

DETAILED DESCRIPTION:
The provision of intraoral palatal anesthesia can be potentially more painful for the patient when compared to other sites of the oral cavity, as palatal tissues are tightly bound to the hard palate with limited tissue space between it and the periosteum . As the injection is given, pressure builds up within the palatal tissues causing pain.

Studies conducted on indirect palatal injection technique (intrapapillary) revealed that it reduces the pain of palatal injection with the same efficacy of anesthesia during extraction.

The desirable method to evade pain during palatal injection is just not to have one. So studies was made to evaluate the single buccal injection and its efficiency during extraction of maxillary teeth. The relatively thin porous bone of posterior buccal maxilla facilitates the diffusion of local anesthetic,as well as articaine can diffuse through soft and hard tissues more reliably than other LA so that maxillary buccal infiltration of articaine provides palatal soft tissue anesthesia.Therefore single injection eliminates the need for multiple painful injections.

ELIGIBILITY:
Inclusion Criteria:

* Children from 6 to 9 years of age requiring extraction in two different quadrants in maxillary arch.

  * Children who demonstrate positive or definitely positive behavior during pretreatment evaluation ranking 3 or 4 in the Frankl scale.

    * Rating 3: Positive Acceptance of treatment; at times cautious; willingness to comply with the dentist, at times with reservation, but patient follows the dentist's directions cooperatively.
    * Rating 4 :Definitely positive Good rapport with the dentists interested in the dental procedures, laughing and enjoying.
  * Child must give assent prior to participation, as well as parental informed written consent.

Exclusion Criteria:

* Medically and mentally compromised children.
* Children with a history of prolonged bleeding, platelet disorders, hypersensitivity,
* History of significant behavior management problems.
* Patients having active sites of pathosis in the area of injection.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Behavior pain assessment during anesthesia and extraction | Intraoperative
  FLACC Behavioral Pain Scale will be used for assessment during anaesthesia and extraction. This scale consists of 5 categories face, leg, activity, cry, consolabilty. Each category is scored on the 0-2 scale, which results in a total score of 0-10.
Subjective self report pain assessment after anesthesia and extraction | intraoperative
  Second subjective self report assesment will be done using Wong-baker scale after the anaesthsia and extraction.It consist of a set of cartoon faces with varying facial expression ranging from smile/laughter to tears.• Each face has a numerical value ranging from 0-5.
physiological record of pain after anesthesia and extraction | intraoperative
  phisiological record including heart rate and blood pressure using an automatic blood pressure monitor.

IPD SHARING:
Plan to Share IPD: Yes
study protocol, informed consent, clinical study report
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After completion of the study
Access Criteria: ClinicalTrials.gov
URL: http://ClinicalTrials.gov